CLINICAL TRIAL: NCT01541488
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Rising Oral Doses (1 mg as Drinking Solution, and 5, 20, 60, 150, 300, 500 mg as Tablets) of BI 1021958 in Healthy Male Volunteers (Placebo-controlled, Randomised and Single Blind Within Dose Groups), Including Investigation of the Effect of Food on the Bioavailability of BI 1021958 (Open-label, Randomised, Two-way Cross-over)
Brief Title: Safety, Tolerability, Pharmacokinetics and Early Pharmacodynamics of Single Rising Oral Doses of BI 1021958 Tablets in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1310.1; 2011-003483-70 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-02-22; First posted 2012-03-01 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Healthy

ARMS (3):
- BI 1021958 (Experimental): Single rising dose (SRD) part
  Interventions: Drug: BI 1021958
- BI 1021958 (Food effect) (Experimental): Food effect part (FE)
  Interventions: Drug: BI 1021958
- Placebo to BI 1021958 (Placebo Comparator): Matching placebo as drinking solution and tablets
  Interventions: Drug: Placebo to BI 1021958

INTERVENTIONS:
Drug: BI 1021958 — tablet
  Arms: BI 1021958 (Food effect)
Drug: BI 1021958 — drinking solution / tablet
  Arms: BI 1021958
Drug: Placebo to BI 1021958 — SRD part: oral administration in fasted state, FE part: oral administration in fasted state and after standard high fat breakfast
  Arms: Placebo to BI 1021958

SUMMARY:
Safety, tolerability, pharmacokinetics and early pharmacodynamics of single rising oral doses of BI 1021958 tablets in healthy male volunteers (first-in-human trial)

ELIGIBILITY:
Inclusion criteria:

1. Healthy male subjects

Exclusion criteria:

1. Any relevant deviation from healthy conditions

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2012-02; Primary Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with clinically relevant findings in physical examination | up to 14 days postdose
Number of participants with clinically relevant findings in vital signs | up to 14 days postdose
Number of participants with clinically significant abnormalities in electrocardiogram (ECG) results | up to 14 days postdose
Number of participants with significant changes from baseline laboratory measurements | up to 14 days postdose
Number of participants with adverse events | up to 14 days postdose
Assessment of tolerability by investigator | up to 14 days postdose

SECONDARY OUTCOMES:
Cmax (maximum measured concentration of BI 1021958 in plasma) | up to 72h postdose
area under the concentration-time curve of BI 1021958 in plasma over the time interval from 0 extrapolated to infinity (AUC0-inf) | up to 72h postdose
AUC0-tz (area under the concentration-time curve of BI 1021958 in plasma over the time interval from 0 up to the last quantifiable data point) | up to 72h postdose

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1310.1.1 Boehringer Ingelheim Investigational Site, Biberach, Germany